CLINICAL TRIAL: NCT07028632
Title: A Phase I/II Study to Assess the Safety, Tolerability and Efficacy of NouvNeu001 Injection for Mid- to Late-stage Parkinson's Disease
Brief Title: The Safety, Feasibility and Efficacy of NouvNeu001 for Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: iRegene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NouvNeu001-02-
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease (PD)
Keywords: Parkinson Disease; Dopaminergic Progenitor Cells
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NouvNeu001 (Experimental)
  Interventions: Biological: Human Dopaminergic Progenitor Cells

INTERVENTIONS:
Biological: Human Dopaminergic Progenitor Cells — Single injection of Human Dopaminergic Progenitor Cells into the putamen/striatum region of brain.

SUMMARY:
This clinical trial is designed to evaluate the safety, tolerability and preliminary efficacy of a single injection of NouvNeu001 (Human Dopaminergic Progenitor Cells Injection) in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This is a multi-center, single arm, and open label trial. The NouvNeu001 will be transplanted into bilateral putamen using stereotactic neurosurgery. Subjects will take immunosuppressants to prevent potential immune rejection for 24 to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years old, male or female
* Able to understand the rationale of the clinical trial and sign informed consent form (ICF)
* Diagnosis of Parkinson's Disease in accordance with the MDS clinical diagnostic criteria for Parkinson's disease (2015)，Parkinson's disease history of ≥ 4 years
* Medically suitable for neurosurgery under anesthesia and able to participate in Computerized Tomography (CT) and Magnetic Resonance Imaging (MRI) and Positron Emission Tomography (PET) scan
* Hoehn-Yahr staging for "off" episodes is 2.5 to 4
* The MDS-UPDRS Part III (MDS-UPDRS-III) score in the "off" state > 35, and positive for the Acute Levodopa Challenge Test (ALCT)
* Currently undergoing treatment with levodopa drugs, but with poor control of motor symptoms or reduced efficacy
* Receive a stable dose of anti-Parkinson's disease drugs for at least 4 weeks before administration
* Acceptable laboratory test results during screening and prior to transplantation
* The patients agreed to postpone any other elective neurosurgery, including deep brain stimulation (DBS), until the completion of the 24-month follow-up
* The patients agreed not to participate in any other interventional clinical studies within 24 months after administration
* The patients agreed not to receive any vaccines within 30 days after administration

Exclusion Criteria:

* Atypical or secondary Parkinson's syndrome to be caused by drugs, metabolic disorders or other reasons
* The patients who have a previous history of PD-related brain surgery and have been judged by the investigator to pose significant risks or impact the assessment, or patients with contraindications for magnetic resonance imaging, or those who have been assessed by the investigator as having any contraindications for surgery or anesthesia, or patients who have received other surgeries that the investigator consider might affect their participation in this study
* There were obvious abnormalities in the cranial CT/MRI examination
* Those who have a history of severe cardiovascular diseases within one year prior to screening
* Patients with a history of malignant tumors，or those who have received cellular therapy or gene therapy within the five years prior to the screening
* Patients with active disseminated intravascular coagulation and significant hemorrhagic tendency within 3 months prior to screening, or who cannot temporarily suspend anti-platelet agents or other anti-coagulant medications for at least 5 days before surgery
* Patients with long-term, heavy use of glucocorticoids or immunosuppressive drugs within 3 months prior to signing the ICF
* Patients with a history of mental illness who are deemed unfit to participate in the study by the investigator; or a history of suicidal ideation or suicide attempts within the past year or currently
* Patients who have used botulinum toxin within 6 months prior to signing the ICF
* Patients with active epilepsy or currently on anti-epileptic drugs
* Patients with a history of dementia or severe cognitive disorder, or the score of MDS-UPDRS 1.1 during screening is > 3; poor compliance, inability to accurately keep diary, and/or inability to sign ICF due to dementia
* Patients with severe depression or with severe anxiety during screening
* Patients with the following abnormalities during screening, including: Abnormal coagulation; Abnormal immunological tests, and assessed by the investigator it is not suitable to participate in the trial; Hypertensive patients with poorly controlled blood pressure and patients with severe postural hypotension; Diabetic patients with poorly controlled blood glucose
* Patients with other combined severe systemic diseases, such as pulmonary heart disease, moderate to severe asthma, severe chronic obstructive pulmonary disease (COPD)
* There are human immunodeficiency virus (HIV) infection, syphilis infection, and active hepatitis C virus (HCV) infection, hepatitis B virus (HBV) infection, tuberculosis infection or other active infections that the investigator consider may affect the participation of the patients in the study or affect the study outcome
* Patients with alcohol addiction or positive for drug of abuse testing
* Patients with a history of contraindication or allergy to the drugs used during the study or any of its components, or are allergic to the same drugs or other macrolides, or have allergies
* Female of childbearing potential who are not surgically sterilized/premenopausal/unwilling to use medically approved effective contraception with 2 years after administration of investigational drug and lactating women; men who are not surgically sterilized/unwilling to use medically approved effective contraception with 2 years after administration of investigational drug
* Patients who have received electric shock therapy within 30 days prior to surgery
* Patients who are participating in other clinical trials, or have been enrolled in other clinical studies and received intervention therapy within 3 months prior to the surgery
* Patients with severe dyskinesia in both on- and off-drug states

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Motor Function | 24 weeks and 48 weeks post-transplant
  Changes in Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part Ⅲ score from baseline to 24 weeks and 48 weeks post-transplant. MDS-UPDRS Part III assesses the motor signs of PD, a higher score indicates more severe symptoms of PD.

SECONDARY OUTCOMES:
The Motor Function and Non-motor Function | 48 weeks and 96 weeks post-transplant
  Changes in MDS-UPDRS Part I-IV Score from baseline to 48 weeks and 96 weeks post-transplant. A higher score indicates more severe symptoms or worse health.
Continued Safety and Tolerability | 96 weeks and 5 years post-transplant
  Incidence and severity of AEs and SAEs within 96 weeks and 5 years post-transplant.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China